CLINICAL TRIAL: NCT03945279
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB100 Administered Orally to Adult Participants With Amyotrophic Lateral Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB100 Administered Orally to Adults With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 261AS101
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: BIIB100 Dose 1 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 2: BIIB100 Dose 2 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 3: BIIB100 Dose 3 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 4: BIIB100 Dose 4 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 5: BIIB100 Dose 5 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 6: BIIB100 Dose 6 (Experimental): Participants will receive single oral dose of BIIB100 on Day 1.
  Interventions: Drug: BIIB100
- Cohort 1-6: Matching Placebo (Placebo Comparator): Participants will receive single oral dose of matching placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB100 — Administered as specified in the treatment arm.
  Arms: Cohort 1: BIIB100 Dose 1; Cohort 2: BIIB100 Dose 2; Cohort 3: BIIB100 Dose 3; Cohort 4: BIIB100 Dose 4; Cohort 5: BIIB100 Dose 5; Cohort 6: BIIB100 Dose 6
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Cohort 1-6: Matching Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability of single-ascending doses of BIIB100 in adults with amyotrophic lateral sclerosis (ALS). The secondary objective of the study is to characterize the pharmacokinetic profile of BIIB100.

ELIGIBILITY:
Key Inclusion Criteria:

* Must meet the laboratory-supported probable, probable, or definite criteria for diagnosing ALS according to the World Federation of Neurology El Escorial criteria.
* Participants taking concomitant riluzole at study entry must be on a stable dose for greater than or equals to (>=) 30 days prior to the first dose of study treatment (Day 1). Participants taking concomitant riluzole must be willing to continue with the same dose regimen throughout the study, unless the Investigator determines that riluzole should be discontinued for medical reasons, in which case it may not be restarted during the study.
* Participants taking concomitant edaravone at study entry must be on a stable dose for >= 60 days prior to the first dose of study treatment (Day 1).
* Adequate respiratory function as indicated by slow vital capacity (SVC) >= 65% of predicted value as adjusted for sex, age, and height (from the sitting position).

Key Exclusion Criteria:

* Ongoing medical condition (e.g., wasting or cachexia, severe anemia) that would, in the opinion of the Investigator, interfere with the conduct or assessments of the study.
* Significant cognitive impairment or unstable psychiatric illness, including psychosis, suicidal ideation, suicide attempt, or untreated major depression less than or equals to (<=) 90 days of Screening, which in the opinion of the Investigator would interfere with the study procedures.
* Treatment with drugs that are transported by Breast Cancer Resistance Protein (BCRP) and P-glycoprotein (P-gp) including, but not limited to, rosuvastatin, sulfasalazine, dabigatran, digoxin and fexofenadine.
* Current enrollment or plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 30 days or 5 half-lives of the agent, whichever is longer, prior to the Baseline Visit (pre-dose on Day 1). Participation in a noninterventional study focused on ALS natural history may be allowed at the discretion of the Investigator and after consultation with the Sponsor.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening (Day -28 ) up to Day 15
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, or is a medically important event.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Maximum Observed Concentration (Cmax) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Time to Reach Cmax (Tmax) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Terminal Elimination Half-life (t1/2) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Apparent Clearance (CL/F) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.
Apparent Volume of Distribution During the Terminal Elimination (Vz/F) of BIIB100 | Day 1 (pre-dose) up to Day 3
  BIIB100 will be measured in the plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (9):
- United States (9):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego Medical Center, San Diego, California
  - Mayo Clinic Hospital, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Johns Hopkins University, Dept of Neurology, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Alliance for Multispecialty Research NOCCR/VRG, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/